CLINICAL TRIAL: NCT02798484
Title: Pilot Study: Monitoring of Breast Cancers Treated by Neoadjuvant Therapy Via Diffusion-weighted Magnetic Resonance Imaging
Brief Title: Monitoring of Breast Cancers Treated by Neoadjuvant Therapy Via Diffusion-weighted Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Mieke Cannie, Head of service, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-CNA
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: Diffusion Weighted Magnetic Resonance Imaging; Breast cancer; Neo-adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast cancer (Experimental): Patients diagnosed with breast cancer and placed under neo-adjuvant treatment (hormonotherapy, chemotherapy) within the CHU Brugmann hospital.
  Interventions: Device: Diffusion-weighted Nuclear Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Diffusion-weighted Nuclear Magnetic Resonance Imaging (MRI) — MRI examinations performed on two devices: Ingernia 3 Testla (Philips) on the Horta site of the CHU Brugmann hospital, and Area 1,5 Tesla (Siemens) on the Brien site of the CHU Brugmann hospital. Diffusion sequences last 6 minutes and are already performed in the standard of care. Compared to the standard of care, one additional MRI will be performed one month after the start of the neo-adjuvant treatment, with diffusion analysis.The post-processing of the examinations will be realized with the Syngo Onco Care application of Siemens.

SUMMARY:
Magnetic resonance imaging (MRI) is the method of choice in breast cancer to perform the loco-regional staging and direct the treatment.

European Guidelines (EUSOMA) currently recommend MRI for initial evaluation and assessement of the neoadjuvant chemotherapy (NAC) response, for breast cancer. The standard of care consists of realizing a MRI before the start of the NAC and another one after it's ended, six months later.

There is currently no consensus on the realization of an interval MRI for early assessment of the chemosensitivity of the tumor. It would allow though alterations in the therapeutic regimen in the event of a non response. Similarly, there is no consensus on when this interval MRI should be performed.

Some recent studies suggest that Diffusion-weighted Magnetic Resonance Imaging is interesting for the evaluation of the early response. However, these are preliminary studies with quantitative measures realized by the region of interest (ROI) method. A response to neoadjuvant chemotherapy results in elevated values of apparent diffusion coefficients (ADC).

The investigator's goal for this study is to evaluate the reliability of diffusion as tumor biomarker. Therefore, they will study the quantitative analysis of the diffusion-weighted magnetic resonance sequences in the pre-therapeutic assessment and the early and late follow-up of breast cancers under neoadjuvant treatment (chemotherapy, hormonotherapy...) within the CHU Brugmann hospital. The results of this analysis will be compared with the MRI results obtained at the end of the treatment and with the histology of the initial biopsy and the surgical specimen.

The expected benefits are:

* to establish correlations between apparent diffusion coefficients (ADC) values and histology
* to observe changes in the ADC according to the type of response: ADC increase in the event of partial response, ADC stability in the event of non response, ADC decrease in the event of a progression, absence of restriction in the event of a complete response.
* to confirm that diffusion weighted MRI within a short interval (after one cure, at one month) has a predictive value for the neoadjuvant chemotherapy (NAC) response.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Neo-adjuvant therapy indication
* Performance status from 0 to 2

Exclusion Criteria:

* Contraindications to magnetic resonance imaging (pacemaker, nerve stimulator, cochlear implant, major claustrophobia)
* Absence of histological results
* Disruption of the neo-adjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Apparent diffusion coefficient (ADC) (mm2/sec) | Baseline: start of the neo-adjuvant therapy
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.
Apparent diffusion coefficient (ADC) (mm2/sec) | One month after the start of the neo-adjuvant therapy
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.
Apparent diffusion coefficient (ADC) (mm2/sec) | At the end of the neo-adjuvant therapy (typical duration: 6 months)
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.
Anatomo-pathology classification - histological type | Baseline: start of the neo-adjuvant therapy
  The histological type of the tumor will be determined by the Anatomo-Pathology Department of the CHU Brugmann hospital, according to standard of care. The determination will be performed on the initial biopsy samples used for diagnosis and/or on the surgical specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Cannie, MD, Principal Investigator — CHU Brugmann; Nathalie Hottat, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Fiorentino C, Berruti A, Bottini A, Bodini M, Brizzi MP, Brunelli A, Marini U, Allevi G, Aguggini S, Tira A, Alquati P, Olivetti L, Dogliotti L. Accuracy of mammography and echography versus clinical palpation in the assessment of response to primary chemotherapy in breast cancer patients with operable disease. Breast Cancer Res Treat. 2001 Sep;69(2):143-51. doi: 10.1023/a:1012277325168. PMID 11759820
- [Background] Vinnicombe SJ, MacVicar AD, Guy RL, Sloane JP, Powles TJ, Knee G, Husband JE. Primary breast cancer: mammographic changes after neoadjuvant chemotherapy, with pathologic correlation. Radiology. 1996 Feb;198(2):333-40. doi: 10.1148/radiology.198.2.8596827.
- [Background] Huber S, Wagner M, Zuna I, Medl M, Czembirek H, Delorme S. Locally advanced breast carcinoma: evaluation of mammography in the prediction of residual disease after induction chemotherapy. Anticancer Res. 2000 Jan-Feb;20(1B):553-8. PMID 10769724
- [Background] Balu-Maestro C, Chapellier C, Bleuse A, Chanalet I, Chauvel C, Largillier R. Imaging in evaluation of response to neoadjuvant breast cancer treatment benefits of MRI. Breast Cancer Res Treat. 2002 Mar;72(2):145-52. doi: 10.1023/a:1014856713942. PMID 12038705
- [Background] Sardanelli F, Boetes C, Borisch B, Decker T, Federico M, Gilbert FJ, Helbich T, Heywang-Kobrunner SH, Kaiser WA, Kerin MJ, Mansel RE, Marotti L, Martincich L, Mauriac L, Meijers-Heijboer H, Orecchia R, Panizza P, Ponti A, Purushotham AD, Regitnig P, Del Turco MR, Thibault F, Wilson R. Magnetic resonance imaging of the breast: recommendations from the EUSOMA working group. Eur J Cancer. 2010 May;46(8):1296-316. doi: 10.1016/j.ejca.2010.02.015. Epub 2010 Mar 19. PMID 20304629
- [Background] Wu LM, Hu JN, Gu HY, Hua J, Chen J, Xu JR. Can diffusion-weighted MR imaging and contrast-enhanced MR imaging precisely evaluate and predict pathological response to neoadjuvant chemotherapy in patients with breast cancer? Breast Cancer Res Treat. 2012 Aug;135(1):17-28. doi: 10.1007/s10549-012-2033-5. Epub 2012 Apr 4. PMID 22476850
- [Background] Li XR, Cheng LQ, Liu M, Zhang YJ, Wang JD, Zhang AL, Song X, Li J, Zheng YQ, Liu L. DW-MRI ADC values can predict treatment response in patients with locally advanced breast cancer undergoing neoadjuvant chemotherapy. Med Oncol. 2012 Jun;29(2):425-31. doi: 10.1007/s12032-011-9842-y. Epub 2011 Feb 1. PMID 21286861
- [Background] Just N. Improving tumour heterogeneity MRI assessment with histograms. Br J Cancer. 2014 Dec 9;111(12):2205-13. doi: 10.1038/bjc.2014.512. Epub 2014 Sep 30. PMID 25268373
- [Derived] Hottat NA, Badr DA, Lecomte S, Besse-Hammer T, Jani JC, Cannie MM. Assessment of diffusion-weighted MRI in predicting response to neoadjuvant chemotherapy in breast cancer patients. Sci Rep. 2023 Jan 12;13(1):614. doi: 10.1038/s41598-023-27787-x. PMID 36635514